CLINICAL TRIAL: NCT06222359
Title: Acceptability of Identifying and Managing Psychological Distress in Multiple Sclerosis: The COMPASS-MS Study
Brief Title: Identifying and Managing Psychological Distress in Multiple Sclerosis: The COMPASS-MS Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 335756
Record Dates: First submitted 2023-11-03; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis; Depression; Anxiety
MeSH Terms: conditions — Multiple Sclerosis; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: COMPASS — Digital CBT to treat psychological distress in Multiple Sclerosis (MS)

SUMMARY:
The aim of this pre-post observational study is to explore if it is feasible to implement 1) routine mental health screening and b) an online Cognitive Behavioural Therapy (CBT) treatment for anxiety and/or depression (named COMPASS-MS) for people living with Multiple Sclerosis (MS) (PwMS) and co-morbid psychological distress in routine care.

DETAILED DESCRIPTION:
The aim of the project is to conduct a feasibility study regarding the implementation of a) routine mental health screening and b) the COMPASS-MS programme as a low-intensity online CBT treatment for anxiety and/or depression in a large English National Health Service (NHS) secondary care MS Clinic.

The intervention will be supported by COMPASS-trained therapists, who will receive supervision from a Clinical Health Psychologist and the Multi-Disciplinary Team (Quantitative Study A). We will also conduct two nested qualitative studies to explore the barriers and facilitators of implementing the COMPASS-MS care pathway locally at King's Hospital (KCH) (Qualitative Study A) and scaling it across Neurology Services outside KCH (Qualitative Study B).

ELIGIBILITY:
Patients will be eligible for inclusion for the COMPASS-MS intervention if they are:

1. Aged ≥18 years
2. Have a diagnosis of MS.
3. Speak English to a sufficiently high standard to allow them to interact with digital CBT programmes.
4. Have access to a computer and email account to allow them to register with the digital CBT programme, and a basic understanding of internet use.
5. Presence of depression and/or anxiety and/or psychological distress evidenced by:

i. A score of ≥ 5 on the nine item self-report measure of depression: PHQ-9 (Kroenke et al., 2001) AND/OR ii. A score of ≥ 5 on the seven item self-report measure of anxiety: GAD-7 (Spitzer et al., 2006).

OR iii. A score of ≥ 10 on the composite measure of depression and anxiety PHQ-ADS (Kroenke et al., 2016).

AND iv. Distress is related to their MS (i.e. answer "yes" or "sometimes" to "Is your distress linked to your MS?"

The below eligibility criteria apply to HCPs who have experience in engaging with COMPASS-MS care pathways at King's College Hospital (KCH).

Healthcare providers (HCPs) will be eligible for inclusion if they meet all or any of the below criteria:

1. Work in the Neurology Service at KCH providing care to PwMS
2. Have experience of either: i) Assessing and triaging patients for psychological distress and/or ii) Providing therapist support to the users of COMPASS-MS.
3. Work in or alongside KCH who are implementing: i) Routine mental health screening ii) COMPASS digital CBT (e.g. pharmacy/physiotherapy commissioning bodies).

Key Stakeholder Inclusion Criteria

Key Stakeholders from Neurology services external to KCH will be invited to take part in an interview if they meet all or any of the below criteria:

1. Work in a Neurology Service in England including both inpatient services and MS therapy centres.
2. Have direct patient experience with working with PwMS (e.g. Neurologist, Doctor, Nurse, Reception)
3. Work alongside a Neurology services in England and are involved in the care of PwMS (e.g. pharmacy/physiotherapy/commissioning bodies).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People living with Multiple Sclerosis (MS) and co-morbid psychological distress Healthcare professionals and Key stakeholders of people living with MS and co-morbid psychological distress
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Psychological Distress (primary outcome for a future full scale trial). | baseline and 12 week follow up
  The investigators will measure general psychological distress using the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS). This includes 9 items from the Patient Health Questionnaire and 7 items from the Generalised Anxiety Disorder Scale. Each item is responded to on a 4-point Likert Scale (0-3) (minimum score: 0, maximum score: 48). Higher scores indicate higher levels of depression and anxiety.

SECONDARY OUTCOMES:
Reach of screening and COMPASS MS intervention | Baseline only
  - The clinical team will collect data on the route of referral to mental health team (completed routine screening, was referred/self-referred).
Reach of screening and COMPASS MS intervention | Baseline only
  - If referred, the clinical team will collect data on the who the referring clinician is and their professional background.
Reach of screening and COMPASS MS intervention | Baseline only
  - The clinical team will collect data on patient attendance at triage appointment and care pathway recommended (including referral to COMPASS-MS)
Reach of screening and COMPASS MS intervention | Baseline only
  - the clinical team will collect data on the outcome of screening (e.g eligible for COMPASS-MS intervention or not)
Efficacy: psychological outcomes | baseline and 12 week follow up
  - The investigators will measure Intolerance of Uncertainty using the Intolerance of Uncertainty Scale-12 item. Items are rated on a 5-point Likert scale (minimum score: 12, maximum score: 60). Higher scores indicate a greater intolerance of uncertainty.
Efficacy: psychological outcomes | baseline and 12 week follow up
  - The investigators will measure Expression of emotion will be measured using the Beliefs about Emotions Scale.
Efficacy: Psycho-social outcomes | baseline and 12 week follow up
  - The investigators will measure Healthcare usage using the 4 service use items from the Client Service Receipt Inventory (CSRI).
Implementation of COMPASS | post treatment (12 week follow up)
  The investigators will investigate the implementation of COMPASS by collecting descriptive data on the number of patients who require digital support to use COMPASS-MS
Implementation of COMPASS | post treatment (12 week follow up)
  The investigators will investigate the implementation of COMPASS by collecting descriptive data on patient adherence to COMPASS online sessions.
Implementation of COMPASS | post treatment (12 week follow up)
  The investigators will investigate the implementation of COMPASS by collecting descriptive data on the number and duration of therapist calls attended.
Implementation of COMPASS | post treatment (12 week follow up)
  The investigators will investigate the implementation of COMPASS by collecting descriptive data on the dropout rate of COMPASS.
Adoption | 12 weeks follow up (post treatment)
  We will qualitatively explore the Adoption of COMPASS.
  We will conduct two nested qualitative studies. 1) we will interview patients and healthcare professionals at Kings College Hospital to explore the barriers and facilitators of implementing the COMPASS-MS care pathway locally at King's Hospital (KCH) (Qualitative Study A) 2 ) we will interview key stakeholders outside of KCH to explore the barriers and facilitators of scaling it across Neurology Services outside KCH (Qualitative Study B).

REFERENCES:
- [Background] Kroenke K, Wu J, Yu Z, Bair MJ, Kean J, Stump T, Monahan PO. Patient Health Questionnaire Anxiety and Depression Scale: Initial Validation in Three Clinical Trials. Psychosom Med. 2016 Jul-Aug;78(6):716-27. doi: 10.1097/PSY.0000000000000322. PMID 27187854
- [Background] Carleton RN, Norton MA, Asmundson GJ. Fearing the unknown: a short version of the Intolerance of Uncertainty Scale. J Anxiety Disord. 2007;21(1):105-17. doi: 10.1016/j.janxdis.2006.03.014. Epub 2006 May 2. PMID 16647833
- [Background] Rimes KA, Chalder T. The Beliefs about Emotions Scale: validity, reliability and sensitivity to change. J Psychosom Res. 2010 Mar;68(3):285-92. doi: 10.1016/j.jpsychores.2009.09.014. Epub 2009 Dec 9. PMID 20159215
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Ryan EG, Vitoratou S, Goldsmith KA, Chalder T. Psychometric Properties and Factor Structure of a Long and Shortened Version of the Cognitive and Behavioural Responses Questionnaire. Psychosom Med. 2018 Feb/Mar;80(2):230-237. doi: 10.1097/PSY.0000000000000536. PMID 29023262
- [Background] Stuifbergen A, Becker H, Blozis S, Beal C. Conceptualization and development of the Acceptance of Chronic Health Conditions Scale. Issues Ment Health Nurs. 2008;29(2):101-14. doi: 10.1080/01612840701792548. PMID 18293219
- [Background] Thornicroft, G. (2001). An adapted version of the Client Service Receipt Inventory. Costing psychiatric interventions. London: Measuring Mental Health Needs.